CLINICAL TRIAL: NCT02190682
Title: Data Collection for Prediction of Postoperative Chronic Pain for Establishing a Software by Using Data Mining Technology
Brief Title: Data Collection for Prediction of Postoperative Chronic Pain for a Software
Status: Completed | Type: Observational
Sponsor: Istanbul University (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Principal Investigator, Prof. Dr. A. Pervin SUTAS BOZKURT, Professor Dr, Istanbul University
Other Study IDs: 2062014
Record Dates: First submitted 2014-07-12; First posted 2014-07-15 (Estimated); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Chronic Postoperative Pain
Keywords: postoperative; chronic; pain; software
MeSH Terms: conditions — Pain, Postoperative; Bronchiolitis Obliterans Syndrome; Pain

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Months
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Postoperative Persistent Pain (PPP) is reported with a high incidence in adults 11.5-47%. This high incidence effects quality of life of patients causes social-economical problems and arises medico-legal issues. This study will be undertaken for producing a database by the evaluation of surgeries in 4 hospitals located in Istanbul. This database will be used in establishing a software by using data mining technology in the prediction of PPP

DETAILED DESCRIPTION:
All cases operated in 4 different hospitals in one month period will be included Exclusion criteria: cases who could not be followed up to 2 months postoperatively by telephone call.

A questionnaire will be filled preoperatively for each case after obtaining informed case . All cases will be anesthetized and pain therapy will be applied according to anesthesiologist's own practice and pain relief will be evaluated and noted. All patients will be telephoned postoperatively for the pain level at 15,30,45 and 60th day. All the information will be uploaded to computer and a software will be prepared for prediction of postoperative chronic pain.

ELIGIBILITY:
Inclusion Criteria:

* all cases operated in one month period

Exclusion Criteria:

* cases who cannot be followed for 2 months

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: all cases undergoing surgery
Sampling Method: Non-Probability Sample
Enrollment: 733 (Actual)
Dates: Start 2014-10 (Actual); Primary Completion 2018-04 (Actual); Study Completion 2018-04-30 (Actual)

PRIMARY OUTCOMES:
Incidence of postoperative chronic pain | postoperative 3 months
  Postoperative chronic pain is pain in the area of surgery lasting at least 2 months postoperatively regardless of infection, recurrence of disease and etc.

SECONDARY OUTCOMES:
preparation of software for the prediction of postoperative chronic pain | 8 months
  the information from the questioners to the patients will be uploaded to an excel sheet and the IT group will prepare a software by using the data mining technology

CONTACTS AND LOCATIONS:
Overall Officials: Pervin Bozkurt Sutaş, Prof. Dr, Study Director — Istanbul University Cerrahpaşa Medical Faculty
Locations (6):
- Turkey (Türkiye) (6):
  - Istanbul University Cerrahpasa Medical Faculty, Istanbul
  - Bezm-i Alem University, Istanbul
  - Istanbul Research and Training Hospital, Istanbul
  - Istanbul University Cardiology Institute, Istanbul
  - Istanbul University Informatics Department, Istanbul
  - Tepecik Research and Training Hospital, Izmir

IPD SHARING:
Plan to Share IPD: Yes
Patient questioner
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Jan 2020- Jan 2022
Access Criteria: when it is published by a journal

REFERENCES:
- [Background] Sutaş Bozkurt, A. P., Özen, Z., Kartal, E., Emre, İ. E., Selçukcan Erol, Ç., Koçoğlu, F. Ö., Güngör, G., Güneyli, H. C., Başaranoğlu, G., Ünlüsoy, E. Ö., Uğur, H. Ö., Buluç Bulğen, S., Çolakoğlu, N., Sayılgan, C., Pekel, A. F., Pişmişoğlu, H., Salihoğlu, Z., Yüceyar, L., Karaca, S., … Bakan, N. (2018). Analysis of the incidence and predictive factors of chronic postoperative pain in adult population. The Journal of Tepecik Education and Research, 28(2), 89-94. https://doi.org/10.5222/terh.2018.089